CLINICAL TRIAL: NCT06886685
Title: Optical Monitoring of Placental Oxygenation and Metabolism
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 156470
Record Dates: First submitted 2025-01-29; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-04

CONDITIONS: Compromised Placental Function
Keywords: pregnant women; fetalsense; fetalsense monitoring; light-based technology; NIRS
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples of whole blood, plasma and serum. Also placenta/cord blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low Risk: Normal pregnancy with fetal gestation of 23 weeks or above
  Interventions: Other: Near Infrared spectroscopy (NIRS)
- High Risk: high-risk pregnancy with fetal gestation of 23 weeks or above with 1 or more of the following issues - hypertensive disorders (including pre-eclampsia (PE), pregnancy induced hypertension and essential hypertension) / pre-existing or gestational diabetes mellitus (GDM) and reactive hypoglycemia (a condition with outcomes similar to GDM according to UCLH research) / Small for Gestational Age (SGA*) / Fetal Growth Restriction (FGR**) and postdates (>40weeks) / with suspected or evidence of infection or inflammation.
  *SGA criteria (as per RCOG GTG 31) - EFW <10th centile.
  ** FGR criteria (as per RCOG GTG 31) - EFW/AC <3rd centile, EFW/AC <10th centile with doppler abnormalities or EFW/AC crossing 2 quartiles on growth charts + doppler abnormalities (CPR<5%/UmA PI >95%).
  Interventions: Other: Near Infrared spectroscopy (NIRS)

INTERVENTIONS:
Other: Near Infrared spectroscopy (NIRS) — NIRS is used as a non-invasive light-based optical technology to measure placental oxygenation and metabolism

SUMMARY:
The aim of this observational study is to detect changes in placental function related to the wellbeing of babies during pregnancy. The study also aims to assess the usefulness of a light-based technology, called near infrared spectroscopy (NIRS), to monitor oxygen levels in the placenta and how placental tissue is using the oxygen (metabolism) during pregnancy.

Participants will be monitored using a newly developed mobile wearable device (light-based technology), which will be placed on the abdomen of pregnant women, and they will be monitored for up to 1 hour during their hospital visit. Participants will attend hospital visits as part of their routine care and these monitoring sessions will take place at this time.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with fetal gestation of 23 weeks or above with:

   * normal or low-risk pregnancy, OR
   * high-risk pregnancy (hypertensive disorders (including preeclampsia (PE), pregnancy induced hypertension and essential hypertension) / pre-existing or gestational diabetes mellitus (GDM) and reactive hypoglycemia (a condition with outcomes similar to GDM according to UCLH research) / Small for Gestational Age (SGA*) / Fetal Growth Restriction (FGR**) and postdates (>40weeks) / with suspected or evidence of infection or inflammation)
2. Singleton Pregnancy
3. Participants aged 18 years or over

   * SGA criteria (as per RCOG GTG 31) - EFW <10th centile. ** FGR criteria (as per RCOG GTG 31) - EFW/AC <3rd centile, EFW/AC <10th centile with doppler abnormalities or EFW/AC crossing 2 quartiles on growth charts + doppler abnormalities (CPR<5%/UmA PI >95%).

Exclusion Criteria:

1. Fetal malformation
2. Fetal genetic and structural abnormalities
3. Participants unable to read and respond to questionnaires in English or Hindi (India)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with fetal gestation of 23 weeks or above
Study Population: Pregnant females aged 18 years old or over.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Compromised placental function and fetal compromise measured by optical instrumentation | through study completion, an average of 6 months
  Assess the relationship between optical markers of oxygenation and metabolism with fetoplacental compromise and outcome. Poor outcomes are defined as Small for Gestational Age (SGA <10th GAP/GROW customised centile) or FGR (fetal growth restriction, defined as EFW or AC <10th centile OR decrease by 50 percentiles17), stillbirth (SB) or poor condition of the newborn infants at birth. Poor condition at birth, fetal death/ death before neonatal hospital discharge, neonatal brain injury syndromes, respiratory support, cardio-vascular abnormality, sepsis and retinopathy of prematurity requiring treatment), while good outcomes indicate live birth of a healthy appropriately grown newborn infant. The primary outcome will be reported with point estimate and corresponding one-sided 95% confidence interval.

SECONDARY OUTCOMES:
Rate of placental oxygenation and metabolism during gestation | through study completion, an average of 6 months
  Develop a monogram of placental oxygenation and metabolism during gestation (23-42 weeks) to characterise the placental development. Investigate the impact of different positions and postures of pregnant women on placental oxygenation.
Association between optical biomarkers and preterm labour | through study completion, an average of 6 months
  Identify proportion of successful monitoring using the optical instrumentation. Combine placental oxygenation, metabolism, fetal heart rate and fetal movement and establish an early warning system for risk identification.
Measure impact of infection and inflammation on placental perfusion and metabolism as well as the newborn brain | through study completion, an average of 6 months
  Associations between optical markers of placental oxygenation and metabolism with placental growth factor (PIGF); placental histological features and gene expression features associated with stillbirth.
Assess impact of fetoplacental compromise on newborn brain and neurodevelopmental follow-up | through study completion, an average of 6 months
  Relationship between optical markers of placental and newborn brain oxygenation and metabolism with neonatal neurodevelopmental follow-up.
Qualitative evaluation of the feasibility and acceptability towards new technology for placental monitoring | through study completion, an average of 9 months
  Interviews at the end of the study to evaluate pregnant women's approach towards the introduction of new technology for placental monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital - UCLH, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No